CLINICAL TRIAL: NCT05613400
Title: The Effect of Simvastatin on Bone Density in Postmenopausal Women With Type 2 Diabetes: a Double-blind, Randomized Active-comparator (Ezetimibe) Controlled Clinical Trial
Brief Title: Statin and Bone Health
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lui Tak Wai David, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STATIN001
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Bone Density; Simvastatin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated 1:1 to 18 months of simvastatin 10mg/day or ezetimibe 10mg/day.
Who Masked: Participant, Investigator
Masking Description: The computer-generated sequence will be supplied by the study statistician, independent of the investigators. To facilitate double-blinding, placebo tablets with the same shapes as simvastatin 10mg and ezetimibe 10mg, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin 10mg/day (Experimental): One simvastatin 10mg-tablet and one placebo tablet with the shape of ezetimibe 10mg each day.
  Interventions: Drug: Simvastatin 10mg
- Ezetimibe 10mg/day (Active Comparator): One ezetimibe 10mg-tablet and one placebo tablet with the shape of simvastatin 10mg each day.
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Simvastatin 10mg — One simvastatin 10mg-tablet
  Arms: Simvastatin 10mg/day
Drug: Ezetimibe 10mg — One ezetimibe 10mg-tablet
  Arms: Ezetimibe 10mg/day

SUMMARY:
This study aims to evaluate the impact of simvastatin on the bone density of postmenopausal women with type 2 diabetes over a duration of 18 months, using a randomized controlled trial design. Aiming to recruit 240 patients, half of them will be randomly assigned to receive simvastatin treatment, while the other half will receive ezetimibe, also a lipid-lowering agent with no known effect on bone. Bone density will be measured at the baseline and the end of the study for comparison of the changes between the simvastatin and the ezetimibe groups.

This is an investigator-initiated study. The principal investigator and the study team will be responsible for ensuring that the study is conducted in compliance with this protocol and the study data collected are verified against the relevant source documents.

All participants will undergo clinical and biochemical assessments at baseline of the trial. Participants will be seen by an endocrinologist at baseline and subsequent follow-up visits at 3, 6, 12 and 18 months respectively.

DETAILED DESCRIPTION:
Study Procedures and Assessments Screening Procedures

Patients will be recruited from medical out-patient clinics, mainly from the primary health care clinics, in the Hong Kong West Cluster of the Hong Kong Hospital Authority. Consecutive participants who fulfil the inclusion and exclusion criteria are invited to participate in this randomized controlled trial after obtaining informed consent.

Clinical and biochemical assessments

Participants will attend a clinical assessment session at baseline after an overnight fast for at least 8 hours. Demographic data and medical history will be obtained using a standardized questionnaire. Personal and family history of fragility fractures (spine, hip, humerus, wrist and ankle) will be recorded. Important clinical risk factors of osteoporosis will be evaluated, including smoking, drinking, family history of fragility fractures, parental history of hip fractures, prior use and duration of hormonal replacement therapy, and levels of physical activity. The levels of physical activity will be assessed through the International Physical Activity Questionnaire (IPAQ). Daily calcium intake will be assessed using a semi-quantitative questionnaire. Body weight, body height and blood pressure (BP) will be measured. Hypertension is defined as BP ≥140/90 mmHg or the use of antihypertensive medications.

Fasting blood will be drawn for plasma glucose, HbA1c, insulin, lipid profile, albumin, calcium, phosphate, creatinine levels and eGFR. Patients with 25OHD levels <50 nmol/L will be given additional cholecalciferol 1000 units/day for 8 weeks followed by reassessment of 25-hydroxyvitamin D (25OHD) to ensure repletion.

Follow-up visits (3, 6, 12, 18 months after baseline visit)

During each follow-up visits, participants will have fasting blood tests checked for liver and renal function tests, creatine kinase, calcium and phosphate, fasting glucose, HbA1c and lipid profile.

Glycaemic control will be managed according to the standard of care. During follow-up visits, tolerance to lipid-lowering therapy will be assessed. Persistent elevation of liver enzymes (alanine aminotransferase and aspartate aminotransferase) to >3 times the upper limit of normal, increase in creatine kinase with clinical signs and symptoms of muscle involvement, or drug intolerance will be excluded from the trial.

During follow-up visits, participants may have changes in clinical conditions and thus be indicated for anti-osteoporosis therapy, or higher-intensity statin. Those who develop incident hip or vertebral fractures, or osteoporosis, and thus require anti-osteoporosis therapy, will be excluded from the trial. Those who develop incident atherosclerotic cardiovascular disease, and thus require higher intensity statin, will also be excluded from the trial.

Withdrawal from study

Patients are informed orally and in writing that they are free to withdraw their participation in the study without bias or prejudice. A patient who decides to stop all therapeutic interventions will be followed by the clinical team for the usual medical care. The date of withdrawal and reason for discontinuation, if known, will be recorded in the medical record.

Statistical Analyses

All statistical analyses will be performed with using R package or IBM® SPSS® version 26. Data will be presented as mean± standard deviation (SD), 95% confidence interval (CI), median with 25th-75th percentile, and number with percentage as appropriate.

All analyses described in this section will be performed based on intention-to-treat analysis and repeated for the per-protocol analysis. Data not normally distributed will be logarithmically transformed before analysis. Between-group comparisons are done with t-test or Mann-Whitney U test for continuous data, and chi-square or Fisher exact test for categorical variables. Two-sided p-value <0.05 will be considered statistically significant.

Baseline demographics and anthropometric parameters (age, BMI), laboratory parameters (HbA1c, LDL-cholesterol, serum creatinine), bone health assessment, including bone mineral density (BMD), trabecular bone score (TBS), bone turnover markers and fracture risk assessment (FRAX) score, clinical risk factors of osteoporosis, family history of fragility fractures (partly reflecting involvement of genetics in bone health), and concomitant medications (various classes of anti-hypertensives and anti-diabetic agents) will be compared between simvastatin and ezetimibe arms.

If applicable, adjustments for covariates may be employed in Analysis of Covariance (ANCOVA). Any adjustments will be pre-specified in the description of the analysis.

BMD is measured with a dual-energy X-ray absorptiometry (DXA) machine (Hologic QDR 4500, Waltham, MA, USA). BMD change over the 18-month period will be calculated for each participant. The BMD change over the lumbar spine (LS), femoral neck (FN), total hip (TH) and distal radius from baseline will be the dependent variable in the ANCOVA model.

Sample size calculation

Sample size calculation is performed with R package (1). According to the study on the impact of lovastatin on TH BMD by Safaei et al. (2), a difference in BMD change over 18-month study period between lovastatin-treated and control groups was 0.098 g/cm2 for TH, with a pooled standard deviation of 0.13 g/cm2. The estimated effect size of TH BMD change over the 18-month study period is 0.75 (95% CI: 0.2-1.3). Assuming the lower CI for the estimated effect size of 0.2, the study would require a sample size of 96 in each group (i.e. total sample size of 192), to achieve 90% power and a level of significance of 5%, for declaring that simvastatin is superior to the active comparator at a 0.02 g/cm2 margin of superiority. To ensure an analysis size of 96 individuals, an overall sample size of 120 individuals per treatment arm will be recruited, anticipating a drop-out rate of approximately 20%.

Protocol Deviations

Protocol deviations are defined as any instance in which the patient or clinical team does not perform scheduled activities/tasks such as missed visits and missed tests and evaluations. Protocols deviations will be reported on the patient's chart.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women
* Aged 50 to 74 years (inclusive);
* Type 2 diabetes Mellitus;
* Postmenopausal: confirmed with the last menstrual period >12 months by the time of recruitment into the study

Exclusion Criteria:

* Entry HbA1c >8.5%;
* On thiazolidinedione;
* Baseline LDL-cholesterol >3.0 mmol/L, triglyceride >5.0 mmol/L, or known familial hypercholesterolaemia;
* History of hip and/or clinical vertebral fractures;
* Osteoporosis by BMD criteria on DXA;
* On anti-osteoporosis therapy within the prior 2 years;
* Evidence of secondary causes of osteoporosis including Cushing's syndrome, acromegaly, thyrotoxicosis, primary hyperparathyroidism, metabolic bone diseases (e.g. osteomalacia), and systemic glucocorticoid treatment;
* Evidence of documented ASCVD, which includes previous acute coronary syndrome, stable angina, coronary revascularization, stroke and transient ischaemic attack and peripheral arterial disease;
* On lipid-lowering therapy within the prior 2 years;
* Known contraindications to statin therapy including allergy, intolerance and significant liver function abnormality (alanine aminotransferase level >3 times upper limit of normal);
* Significant diabetic complication(s): pre-proliferative / proliferative diabetic retinopathy, diabetic maculopathy, overt proteinuria, estimated glomerular filtration rate (eGFR) <30 mL/min;
* Inability to give an informed consent

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The change in the TH BMD after 18 months of simvastatin compared with ezetimibe | Screening visit and Visit 5 (18 month after baseline visit)
  BMD at the TH will be measured with DXA and compared.

SECONDARY OUTCOMES:
The changes in the LS BMD after 18 months of simvastatin compared with ezetimibe | Screening visit and Visit 5 (18 month after baseline visit)
  BMD at the LS will be measured with DXA and compared.
The changes in the FN BMD after 18 months of simvastatin compared with ezetimibe | Screening visit and Visit 5 (18 month after baseline visit)
  BMD at the FN will be measured with DXA and compared.
The changes in BMD over distal radius after 18 months of simvastatin compared with ezetimibe | Screening visit and Visit 5 (18 month after baseline visit)
  BMD at the distal radius will be measured with DXA and compared.
The changes in bone turnover marker, carboxy-terminal cross-linked telopeptide of type 1 collagen (CTX) after 6 months and 18 months of simvastatin compared with ezetimibe | Baseline visit, Visit 3 (6 months after Baseline visit) and Visit 5 (18 months after Baseline visit)
The changes in bone turnover marker, amino-terminal propeptides of type 1 collagen (P1NP) after 6 months and 18 months of simvastatin compared with ezetimibe | Baseline visit, Visit 3 (6 months after Baseline visit) and Visit 5 (18 months after Baseline visit)
The changes in TBS after 18 months of simvastatin compared with ezetimibe | Screening visit and Visit 5 (18 month after baseline visit)
  A higher TBS indicates better quality of bone which is less likely to fracture. The minimum value of TBS is 0.8, while the maximum value of TBS is 1.6.

CONTACTS AND LOCATIONS:
Overall Officials: Tak Wai David Lui, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Diabetes Centre, 2/F, Block L, Department of Medicine, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. 2008. 58 p.
- [Background] Safaei H, Janghorbani M, Aminorroaya A, Amini M. Lovastatin effects on bone mineral density in postmenopausal women with type 2 diabetes mellitus. Acta Diabetol. 2007 Jun;44(2):76-82. doi: 10.1007/s00592-007-0246-6. Epub 2007 May 27. PMID 17530471
- [Background] Pisani P, Renna MD, Conversano F, Casciaro E, Di Paola M, Quarta E, Muratore M, Casciaro S. Major osteoporotic fragility fractures: Risk factor updates and societal impact. World J Orthop. 2016 Mar 18;7(3):171-81. doi: 10.5312/wjo.v7.i3.171. eCollection 2016 Mar 18. PMID 27004165
- [Background] Tatangelo G, Watts J, Lim K, Connaughton C, Abimanyi-Ochom J, Borgstrom F, Nicholson GC, Shore-Lorenti C, Stuart AL, Iuliano-Burns S, Seeman E, Prince R, March L, Cross M, Winzenberg T, Laslett LL, Duque G, Ebeling PR, Sanders KM. The Cost of Osteoporosis, Osteopenia, and Associated Fractures in Australia in 2017. J Bone Miner Res. 2019 Apr;34(4):616-625. doi: 10.1002/jbmr.3640. Epub 2019 Jan 7. PMID 30615801
- [Background] Lee PCH, Woo YC, Lam KSL. Fighting the Health Challenges of Diabetes in Hong Kong: A Window Into Mainland China. Am J Public Health. 2018 Dec;108(12):1623-1624. doi: 10.2105/AJPH.2018.304740. No abstract available. PMID 30403505
- [Background] 55th EASD Annual Meeting of the European Association for the Study of Diabetes : Barcelona, Spain, 16 - 20 September 2019. Diabetologia. 2019 Sep;62(Suppl 1):1-600. doi: 10.1007/s00125-019-4946-6. No abstract available. PMID 31384961
- [Background] Ma L, Oei L, Jiang L, Estrada K, Chen H, Wang Z, Yu Q, Zillikens MC, Gao X, Rivadeneira F. Association between bone mineral density and type 2 diabetes mellitus: a meta-analysis of observational studies. Eur J Epidemiol. 2012 May;27(5):319-32. doi: 10.1007/s10654-012-9674-x. Epub 2012 Mar 27. PMID 22451239
- [Background] Janghorbani M, Van Dam RM, Willett WC, Hu FB. Systematic review of type 1 and type 2 diabetes mellitus and risk of fracture. Am J Epidemiol. 2007 Sep 1;166(5):495-505. doi: 10.1093/aje/kwm106. Epub 2007 Jun 16. PMID 17575306
- [Background] Lui DTW, Lee CH, Chan YH, Chow WS, Fong CHY, Siu DCW, Tse HF, Woo YC, Lam KSL. HbA1c variability, in addition to mean HbA1c, predicts incident hip fractures in Chinese people with type 2 diabetes. Osteoporos Int. 2020 Oct;31(10):1955-1964. doi: 10.1007/s00198-020-05395-z. Epub 2020 May 8. PMID 32385660
- [Background] Liao CC, Lin CS, Shih CC, Yeh CC, Chang YC, Lee YW, Chen TL. Increased risk of fracture and postfracture adverse events in patients with diabetes: two nationwide population-based retrospective cohort studies. Diabetes Care. 2014 Aug;37(8):2246-52. doi: 10.2337/dc13-2957. Epub 2014 May 7. PMID 24804698
- [Background] Yun-Ning Cheung E, Pik-Shan Kong A, Siu-Him Lau E, Yee-Kwan Chow E, On-Yan Luk A, Ching-Wan Ma R, Ping Lam T, Yuk-Wai Lee W, Chun-Yiu Cheng J, Ebeling PR, Chung-Ngor Chan J. Association of hip fractures with cardiometabolic-renal risk factors in Southern Chinese patients with type 2 diabetes - the Hong Kong Diabetes Register. J Diabetes Investig. 2021 Sep;12(9):1739-1748. doi: 10.1111/jdi.13529. Epub 2021 Mar 15. PMID 33605046
- [Background] Lecka-Czernik B. Diabetes, bone and glucose-lowering agents: basic biology. Diabetologia. 2017 Jul;60(7):1163-1169. doi: 10.1007/s00125-017-4269-4. Epub 2017 Apr 22. PMID 28434032
- [Background] Leslie WD, Aubry-Rozier B, Lamy O, Hans D; Manitoba Bone Density Program. TBS (trabecular bone score) and diabetes-related fracture risk. J Clin Endocrinol Metab. 2013 Feb;98(2):602-9. doi: 10.1210/jc.2012-3118. Epub 2013 Jan 22. PMID 23341489
- [Background] Karlson BW, Palmer MK, Nicholls SJ, Lundman P, Barter PJ. A VOYAGER Meta-Analysis of the Impact of Statin Therapy on Low-Density Lipoprotein Cholesterol and Triglyceride Levels in Patients With Hypertriglyceridemia. Am J Cardiol. 2016 May 1;117(9):1444-8. doi: 10.1016/j.amjcard.2016.02.011. Epub 2016 Feb 17. PMID 26969416
- [Background] Ferrari SL, Abrahamsen B, Napoli N, Akesson K, Chandran M, Eastell R, El-Hajj Fuleihan G, Josse R, Kendler DL, Kraenzlin M, Suzuki A, Pierroz DD, Schwartz AV, Leslie WD; Bone and Diabetes Working Group of IOF. Diagnosis and management of bone fragility in diabetes: an emerging challenge. Osteoporos Int. 2018 Dec;29(12):2585-2596. doi: 10.1007/s00198-018-4650-2. Epub 2018 Jul 31. PMID 30066131
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Man LP, Ho AW, Wong SH. Excess mortality for operated geriatric hip fracture in Hong Kong. Hong Kong Med J. 2016 Feb;22(1):6-10. doi: 10.12809/hkmj154568. Epub 2015 Oct 9. PMID 26494900
- [Background] Authors/Task Force Members; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2019 ESC/EAS guidelines for the management of dyslipidaemias: Lipid modification to reduce cardiovascular risk. Atherosclerosis. 2019 Nov;290:140-205. doi: 10.1016/j.atherosclerosis.2019.08.014. Epub 2019 Aug 31. No abstract available. PMID 31591002
- [Background] Oryan A, Kamali A, Moshiri A. Potential mechanisms and applications of statins on osteogenesis: Current modalities, conflicts and future directions. J Control Release. 2015 Oct 10;215:12-24. doi: 10.1016/j.jconrel.2015.07.022. Epub 2015 Jul 28. PMID 26226345
- [Background] Moon HJ, Kim SE, Yun YP, Hwang YS, Bang JB, Park JH, Kwon IK. Simvastatin inhibits osteoclast differentiation by scavenging reactive oxygen species. Exp Mol Med. 2011 Nov 30;43(11):605-12. doi: 10.3858/emm.2011.43.11.067. PMID 21832867
- [Background] Chung YS, Lee MD, Lee SK, Kim HM, Fitzpatrick LA. HMG-CoA reductase inhibitors increase BMD in type 2 diabetes mellitus patients. J Clin Endocrinol Metab. 2000 Mar;85(3):1137-42. doi: 10.1210/jcem.85.3.6476. PMID 10720052
- [Background] Nakashima A, Nakashima R, Ito T, Masaki T, Yorioka N. HMG-CoA reductase inhibitors prevent bone loss in patients with Type 2 diabetes mellitus. Diabet Med. 2004 Sep;21(9):1020-4. doi: 10.1111/j.1464-5491.2004.01292.x. PMID 15317608
- [Background] Bouxsein ML, Eastell R, Lui LY, Wu LA, de Papp AE, Grauer A, Marin F, Cauley JA, Bauer DC, Black DM; FNIH Bone Quality Project. Change in Bone Density and Reduction in Fracture Risk: A Meta-Regression of Published Trials. J Bone Miner Res. 2019 Apr;34(4):632-642. doi: 10.1002/jbmr.3641. Epub 2019 Jan 23. PMID 30674078
- [Background] Graham DJ, Staffa JA, Shatin D, Andrade SE, Schech SD, La Grenade L, Gurwitz JH, Chan KA, Goodman MJ, Platt R. Incidence of hospitalized rhabdomyolysis in patients treated with lipid-lowering drugs. JAMA. 2004 Dec 1;292(21):2585-90. doi: 10.1001/jama.292.21.2585. Epub 2004 Nov 22. PMID 15572716
- [Background] Charles EC, Olson KL, Sandhoff BG, McClure DL, Merenich JA. Evaluation of cases of severe statin-related transaminitis within a large health maintenance organization. Am J Med. 2005 Jun;118(6):618-24. doi: 10.1016/j.amjmed.2005.02.008. PMID 15922693
- [Background] Knopp RH, Gitter H, Truitt T, Bays H, Manion CV, Lipka LJ, LeBeaut AP, Suresh R, Yang B, Veltri EP; Ezetimibe Study Group. Effects of ezetimibe, a new cholesterol absorption inhibitor, on plasma lipids in patients with primary hypercholesterolemia. Eur Heart J. 2003 Apr;24(8):729-41. doi: 10.1016/s0195-668x(02)00807-2. PMID 12713767
- [Background] Mei J, Yeung SS, Kung AW. High dietary phytoestrogen intake is associated with higher bone mineral density in postmenopausal but not premenopausal women. J Clin Endocrinol Metab. 2001 Nov;86(11):5217-21. doi: 10.1210/jcem.86.11.8040. PMID 11701680
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462

DOCUMENTS (2):
  • Study Protocol (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05613400/Prot_000.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05613400/ICF_001.pdf